CLINICAL TRIAL: NCT02540083
Title: Assessment of Diagnostic Accuracy and Performance of Digital Breast Tomosynthesis Compared to Mammography ADAPT-Enrich: Recruitment Plan for Initially Asymptomatic Women Referred for Breast Biopsy After Screening Digital Breast Tomosynthesis Exam
Brief Title: Assessment of Diagnostic Accuracy and Performance of Digital Breast Tomosynthesis Compared to Mammography
Acronym: ADAPT-ENRICH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor has obtained sufficient case load prematurely.
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 124.03-2015-GES-0001
Record Dates: First submitted 2015-09-01; First posted 2015-09-03 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Breast Cancer; Tumors, Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental: DBT and FFDM (Experimental): Subjects underwent 2D breast imaging with full-field digital mammography (FFDM) followed by 3D breast imaging with digital breast tomosynthesis (DBT).
  Interventions: Device: DBT and FFDM

INTERVENTIONS:
Device: DBT and FFDM — Subjects underwent FFDM breast imaging followed by DBT breast imaging
  Other Names: Digital Breast Tomosynthesis (3D breast imaging) DBT; Full-Field Digital Mammography (2D breast imaging) FFDM

SUMMARY:
The aim of this recruitment plan (ADAPT-Enrich) is to collect image and technical data on both digital breast tomosynthesis (DBT) and full-field digital mammography (FFDM), along with other subject data including histology results from biopsy specimen examination and cancer classification data from initially asymptomatic women referred for clinically indicated breast biopsy based on suspicious DBT screening breast imaging results. These data will be included in a subsequent and prospectively planned pooled analysis described in a separate protocol (ADAPT-BIE) examining superiority of DBT to FFDM for breast cancer diagnosis and other performance measures.

DETAILED DESCRIPTION:
ADAPT-ENRICH will supplement an on-going program (ADAPT) which consists of 2 additional recruitment plans (ADAPT-SCR and ADAPT-BX) followed by an off-line read of the images and data collected (ADAPT-BIE). This study involves the comparison of two devices that can identify abnormalities in routine breast screening and diagnostic mammography. Mammography is usually done with full-field digital mammography (FFDM), which takes flat, two-dimensional X-ray images of the breast. Doctors use the two-dimensional images to look for cancers and other abnormal tissue. The purpose of this study is to learn more about the accuracy of full-field digital mammography devices and a new mammography device called digital breast tomosynthesis (DBT). DBT is similar to full-field digital mammography, but can also move around the breast to get X-ray images from different angles, which provides a three-dimensional view that doctors can use to look for cancers and abnormal tissue. Subjects will be recruited from an initially asymptomatic population that have been referred for clinically indicated breast biopsy based on suspicious DBT screening breast imaging results. Subjects will undergo a DBT mammogram prior to biopsy. If FFDM was not performed within 30 days, subjects will also undergo FFDM prior to biopsy. Results of biopsy(ies) and histopathology, including lesion characteristics, will be recorded and considered as truth if positive for cancer status. Subjects with negative or benign histological findings will be followed for approximately one year (10-16 months) by FFDM and any additional standard of care practice.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 30 years or older (≥30 years old);
* Initially asymptomatic women who underwent routine bilateral screening with Digital Breast Tomosynthesis (DBT), followed by diagnostic work-up showing one or more abnormalities and referred for breast biopsy;
* Are able and willing to comply with study procedures;
* Have signed and dated the informed consent form;
* Documented as non-pregnant based on the investigator's medical judgment and in consideration of local clinical practice standards for evidence of non-pregnancy.

Exclusion Criteria:

* Have been previously included in this study , ADAPT-SCR recruitment plan or ADAPT-BX recruitment plan;
* Have undergone diagnostic or surgical intervention(s) or procedure(s) on either breast, including mastectomy and cytopunction, before study-related imaging;
* Have breasts too large to be adequately positioned on 24 x 31 centimeter (cm) DBT or FFDM digital receptor without anatomical cut-off during a DBT or FFDM examination;
* Have participated in (within the prior 30 days) another trial of an investigational product expected to interfere with study procedures or outcomes;
* Have breast implant(s);
* Have reconstructed breast(s).

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Carolina Breast Imaging Specialists, Greenville, North Carolina
  - Avera Breast Center, Sioux Falls, South Dakota

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental: DBT and FFDM
Started | 94
Completed | 78
Not Completed | 16
Not completed — Withdrawal by Subject | 16

BASELINE CHARACTERISTICS:
Population: Population includes study participants who completed DBT, FFDM and lesion biopsy.
Arm/Group | Experimental: DBT and FFDM
Number analyzed (Participants) | 78
Age, Continuous [Mean (Full Range); unit: years] | 52.8 [31 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 78

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With DBT, FFDM and Biopsy Specimens Collected
Description: For each participant, obtain image data using two methods (DBT and FFDM) and obtain histology results of biopsy specimens from women referred for biopsy.
Time Frame: Approximately 8 weeks
Population: Total number of participants enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: DBT and FFDM
Number analyzed (Participants) | 94
Participants
  Participants that completed DBT, FFDM and Biopsy | 78
  Participants taht did not complete all three tests | 16

2. Secondary Outcome: Lesion Type Observed by FFDM Imaging
Description: Lesions were characterized based on findings identified during image evaluations performed by qualified readers.
Time Frame: Approximately 8 weeks
Population: Lesions observed using FFDM imaging
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Experimental: DBT and FFDM
Number analyzed (Participants) | 78
Number analyzed (Lesions) | 107
Lesions
  Lesion type = mass | 43
  Lesion type = calcification | 32
  Lesion type = all other | 32

3. Secondary Outcome: Lesion Type Observed by DBT Imaging
Description: Lesions were characterized based on findings identified during image evaluations performed by qualified researchers.
Time Frame: Approximately 8 weeks
Population: Lesions observed using DBT
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Experimental: DBT and FFDM
Number analyzed (Participants) | 78
Number analyzed (lesions) | 118
lesions
  Lesion description = mass | 51
  Lesion description = calcification | 33
  Lesion description = all other | 34

4. Secondary Outcome: Lesion Size as Observed by FFDM
Description: Length of Lesions (measured in mm) when images were collected using FFDM.
Time Frame: Approximately 8 weeks
Population: Lesions as observed by FFDM
Measure: Mean (Full Range); unit: millimeters (mm)
Units Other Than Participants: Lesions
Arm/Group | Experimental: DBT and FFDM
Number analyzed (Participants) | 78
Number analyzed (Lesions) | 88
millimeters (mm) | 15.3 [3.0 to 80.0]

5. Secondary Outcome: Lesion Size as Observed by DBT
Description: Length of lesions (measured in mm) when images were collected using DBT.
Time Frame: Approximately 8 weeks
Population: Lesions observed and measured when images were collected using DBT
Measure: Mean (Full Range); unit: millimeters (mm)
Units Other Than Participants: lesions
Arm/Group | Experimental: DBT and FFDM
Number analyzed (Participants) | 78
Number analyzed (lesions) | 111
millimeters (mm) | 13.8 [1.5 to 66.0]

6. Secondary Outcome: Biopsy Finding of Lesions
Description: Describes histologic cancer and non-cancer findings of lesion biopsy.
Time Frame: Approximately 8 weeks
Population: All participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: DBT and FFDM
Number analyzed (Participants) | 78
Participants
  Lesion is "positive/malignant" | 32
  Lesion is "negative/benign" | 43
  Biopsy was non-conclusive | 3

7. Other Pre Specified Outcome: Safety - Device Related Malfunctions
Description: Number of device-related malfunctions by imaging modality.
Time Frame: Approximately 8 weeks
Population: All enrolled participants
Measure: Number; unit: malfunctions
Arm/Group | Experimental: DBT and FFDM
Number analyzed (Participants) | 94
malfunctions
  Device malfunctions for FFDM | 0
  Device malfunctions for DBT | 0

ADVERSE EVENTS:
Time Frame: AE data was collected for each subject for the duration that they were on site for DBT or FFDM scans. For all subjects, duration of study was approximately 21 months.
Arm/Group | Experimental: DBT and FFDM
All-Cause Mortality (participants affected / at risk) | 0/94
Serious Adverse Events (participants affected / at risk) | 0/94
Other Adverse Events (participants affected / at risk) | 0/94

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-23): https://cdn.clinicaltrials.gov/large-docs/83/NCT02540083/Prot_SAP_000.pdf